CLINICAL TRIAL: NCT00218868
Title: Cytodiagnosis of Basal Cell Carcinoma and Actinic Keratosis Using Papanicolaou and May-grunvald-giemsa Stained Cutaneous Tissue Smear in Relation to Photodynamic Therapy
Brief Title: Cytodiagnosis of Basal Cell Carcinoma and Actinic Keratosis Using Papanicolaou and May-grunwald-giemsa Stained Tissue Smear
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: EC-001
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Carcinoma, Basal Cell; Porokeratosis, Disseminated Superficial Actinic
Keywords: Cytodiagnosis; Skin Scrape; Touch Imprint; Papanicolaou; May-Grunvald-Giemsa
MeSH Terms: conditions — Carcinoma, Basal Cell; Porokeratosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- skin scrape
  Interventions: Procedure: Skin scrape

INTERVENTIONS:
Procedure: Skin scrape — scrape cytology using two different cytological staining techniques, and additional touch imprint cytology compared with histopathology of superficial basal cell carcinoma and actinic keratosis

SUMMARY:
The purpose of this study is to compare and evaluate the diagnostic performance of scrape cytology using two different cytological staining techniques, and to evaluate additional touch imprint cytology with that of histopathology of superficial basal cell carcinoma and actinic keratosis.

ELIGIBILITY:
Inclusion Criteria:

Histologically verified basal call carcinoma and actinic keratosis

Exclusion Criteria:

Morphea form of basal cell carcinoma. Pigmented form of basal cell carcinoma.

Ages: 0 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 50 BCC and 28 AK histologically verified lesions, from 41 and 25 patients, respectively
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2000-01; Primary Completion 2006-02 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eidi Christensen, MD, Principal Investigator — St. Olav, University Hospital, Trondheim
Locations (1):
- St. Olav University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Christensen E, Bofin A, Gudmundsdottir I, Skogvoll E. Cytological diagnosis of basal cell carcinoma and actinic keratosis, using Papanicolaou and May-Grunwald-Giemsa stained cutaneous tissue smear. Cytopathology. 2008 Oct;19(5):316-22. doi: 10.1111/j.1365-2303.2007.00483.x. Epub 2007 Oct 4. PMID 17916094